CLINICAL TRIAL: NCT04826588
Title: Randomised Evaluation of COVID-19 Therapy (RECOVERY) in Children With PIMS-TS in Switzerland (SWISSPED-RECOVERY)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Collaborators: SwissPedNet (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-00362; ks21Bielicki2
Record Dates: First submitted 2021-03-31; First posted 2021-04-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2023-02

CONDITIONS: Paediatric Inflammatory Multisystem Syndrome-Temporally Associated With SARS-CoV-2 (PIMS-TS)
Keywords: coronavirus-disease (COVID-19); SARS coronavirus 2 (SARS-CoV-2); tocilizumab; anakinra; Human normal immunoglobulin (IVIg); Methylprednisolone sodium succinate
MeSH Terms: conditions — pediatric multisystem inflammatory disease, COVID-19 related; COVID-19 | interventions — Methylprednisolone Hemisuccinate; gamma-Globulins; Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: Overarching trial design with treatment arms that are both available at the hospital and not believed by the enrolling doctor to be contraindicated (e.g. by particular co-morbid conditions or concomitant medications). Treatment arms to be added or removed according to the emerging evidence.
  Main randomisation part A: Methylprednisolone 2 mg/kg for three days intravenous or orally vs corticosteroids methylprednisolone 10mg/kg intravenous for three days vs intravenous immunoglobulin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone sodium succinate 10 mg/kg (Active Comparator): Methylprednisolone sodium succinate 10 mg/kg intravenously once daily for 3 days (max 1 g per dose)
  Interventions: Drug: Methylprednisolone sodium succinate 10 mg/kg intravenously
- Human normal immunoglobulin (IVIg) (Active Comparator): Human normal immunoglobulin (IVIg) 2g/kg intravenously as a single dose in line with guidance for dosing and administration in Kawasaki disease
  Interventions: Biological: Human normal immunoglobulin (IVIg)

INTERVENTIONS:
Drug: Methylprednisolone sodium succinate 10 mg/kg intravenously — Methylprednisolone sodium succinate 10 mg/kg intravenously once daily for 3 days (max 1 g per dose)
  Arms: Methylprednisolone sodium succinate 10 mg/kg
Biological: Human normal immunoglobulin (IVIg) — Human normal immunoglobulin (IVIg) 2g/kg intravenously as a single dose in line with guidance for dosing and administration in Kawasaki disease
  Arms: Human normal immunoglobulin (IVIg)

SUMMARY:
The study is to provide reliable estimates of the effect of study treatment on hospital length of stay through to 28 days after randomisation.

The protocol describes an overarching trial design to provide reliable evidence on the efficacy of candidate therapies for children hospitalised with PIMS-TS. It is an adaptive pragmatic platform trial with an open-label randomisation.

New trial arms can be added as evidence emerges that other candidate therapeutics should be evaluated.

DETAILED DESCRIPTION:
In May 2020 a new COVID-associated inflammatory syndrome in children was identified, Paediatric Inflammatory Multisystem Syndrome - Temporally associated with SARS-CoV-2 (PIMS-TS). A rapid international consensus process identified the need to evaluate corticosteroids and intravenous immunoglobulin (IVIg) as initial therapies in PIMS-TS, and confirmed tocilizumab and anakinra as biological anti-inflammatory agents to be evaluated as a second line therapy.

This Swissped-Recovery trial is a sister trial to the RECOVERY international trial with the implementation of the study at Swiss study sites.

The protocol describes an overarching trial design to provide reliable evidence on the efficacy of candidate therapies for children hospitalised with PIMS-TS. It is an adaptive pragmatic platform trial with an open-label randomisation.

New trial arms can be added as evidence emerges that other candidate therapeutics should be evaluated.

Additional substudies can be added to provide more detailed information on side effects or sub-categorisation of patient types.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised children (aged <18 years old)
* SARS-CoV-2 infection associated disease (clinically suspected or laboratory confirmed) with evidence of single or multi-organ dysfunction (called Pediatric Multisystem Inflammatory Syndrome temporally associated with COVID-19 [PIMS-TS]).
* No medical history that might, in the opinion of the attending clinician, put the patient at significant risk if he/she were to participate in the trial

Exclusion Criteria:

* Neonates/infants with a corrected gestational age of <= 44 weeks
* If the attending clinician believes that there is a specific contra-indication to one of the active drug treatment arms or that the patient should definitely be receiving one of the active drug treatment arms, then that arm will not be available for randomisation for that patient.

Ages: 44 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2021-05-23 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | Within 28 days after randomisation
  effect of study treatment on hospital length of stay

SECONDARY OUTCOMES:
All-cause mortality among patients | Within 28 days and up to 6 months after randomisation
  For each pairwise comparison with the 'no additional treatment' arm, the primary objective is to provide reliable estimates of the effect of study treatments on all-cause mortality.
Composite endpoint of death or need for mechanical ventilation or extracorporeal membrane oxygenation (ECMO) | Within 28 days and up to 6 months after randomisation
  Among patients not on invasive mechanical ventilation at baseline, the number of patients with a composite endpoint of death or need for invasive mechanical ventilation or ECMO.

OTHER OUTCOMES:
Need for (and duration of) ventilation | Within 28 days and up to 6 months after randomisation
  To assess the effects of study treatment on number of patients who needed any ventilation and (for invasive mechanical ventilation) the number of days it was required
Need for renal replacement therapy | Within 28 days and up to 6 months after randomisation
  To assess the effects of study treatment on number of patients who needed renal replacement therapy
Number of patients who had thrombotic events | Within 28 days and up to 6 months after randomisation
  To assess the effects of study treatment on number of patients who had thrombotic events
Cardiac outcome (long-term impact) of PIMS-TS after discharge | Post-discharge extended follow-up visits up to 6 months after randomisation
  Cardiac function and presence of coronary artery aneurysms will be assessed by echocardiography.
Neurological outcome (long-term impact) of PIMS-TS after discharge | Post-discharge extended follow-up visits up to 6 months after randomisation
  assessment of post-traumatic stress disorder
Health care costs | Within 28 days after randomisation
  Direct hospitalization-related costs will be captured for health economic analyses. For each PIMS-TS related hospitalization episode recruited in the study, the total Diagnosis-Related Group (DRG) costs claimed by the respective study site will be extracted from the institutional finance records, and analysed in batch upon completion of recruitment
Quality of life post-infection assessed by Strengths and Difficulties Questionnaire (SDQ) | Post-discharge extended follow-up visits up to 6 months after randomisation
  The strengths and difficulties questionnaire (SDQ) is a short behavioural screening questionnaire for children aged 3 to 16. The 25 personality attributes in the SDQ are made up of 5 scales of 5 items each. The scales are:
  Emotional symptoms, Conduct problems, Hyperactivity/inattention, Peer relationship problems, Prosocial behaviour. Each subscale includes five items, rating each item as either: Never = 0, Somewhat True = 1 or Certainly True = 2. SDQ total scores of 17 and above are considered to be abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Bielicki, Dr. med., Principal Investigator — Paediatric Infectious Diseases and Vaccinology, Universität-Kinderspital beider Basel (UKBB); Luregn Schlapbach, Dr. med., Principal Investigator — Pediatric and Neonatal Intensive Care Unit, University Children's Hospital Zurich
Locations (10):
- Switzerland (10):
  - Cantonal Hospital Aarau, Department of Paediatrics, Aarau
  - University of Basel Children's Hospital, Basel
  - Ente Ospedaliero Cantonale Ticino (EOC) Pediatrica, Bellinzona
  - Department of Pediatrics, University of Bern, Bern
  - Department of Child, Woman and, Adolescent Medecine, Geneva University Hospitals and Faculty of Medicine, Geneva
  - Department of Pediatrics,University Hospital of Lausanne (CHUV), Lausanne
  - Department of Pediatrics, Cantonal Hospital Luzern, Lucerne
  - Children's Hospital of Eastern Switzerland, Sankt Gallen
  - Department of Pediatrics, Cantonal Hospital Fribourg, Villars-sur-Glâne
  - University Children's Hospital Zuerich, Zurich

REFERENCES:
- [Result] Welzel T, Atkinson A, Schobi N, Andre MC, Bailey DGN, Blanchard-Rohner G, Buettcher M, Grazioli S, Koehler H, Perez MH, Truck J, Vanoni F, Zimmermann P, Sanchez C, Bielicki JA, Schlapbach LJ; Swissped RECOVERY Trial Group. Methylprednisolone versus intravenous immunoglobulins in children with paediatric inflammatory multisystem syndrome temporally associated with SARS-CoV-2 (PIMS-TS): an open-label, multicentre, randomised trial. Lancet Child Adolesc Health. 2023 Apr;7(4):238-248. doi: 10.1016/S2352-4642(23)00020-2. Epub 2023 Feb 3. PMID 36746174
- [Derived] Schobi N, Sanchez C, Welzel T, Bamford A, Webb K, Rojo P, Tremoulet A, Atkinson A, Schlapbach LJ, Bielicki JA; Swissped-RECOVERY trial group. Swissped-RECOVERY: masked independent adjudication for the interpretation of non-randomised treatment in a two-arm open-label randomised controlled trial (methylprednisolone vs immunoglobulins) in Paediatric Inflammatory Multisystem Syndrome Temporally Associated with SARS-CoV-2 (PIMS-TS) involving 10 secondary and tertiary paediatric hospitals in Switzerland. BMJ Open. 2024 Apr 25;14(4):e078137. doi: 10.1136/bmjopen-2023-078137. PMID 38670610
- [Derived] Andre MC, Sanchez C, Bressieux-Degueldre S, Perez MH, Wutz D, Blanchard-Rohner G, Grazioli S, Schobi N, Truck J, Welzel T, Atkinson A, Schlapbach LJ, Bielicki J; Swissped RECOVERY Trial Group. Cardiac assessment and inflammatory markers in children with paediatric inflammatory multisystem syndrome temporally associated with SARS-CoV2 (PIMS-TS) treated with methylprednisolone versus intravenous immunoglobulins: 6-month follow-up outcomes of the randomised controlled Swissped RECOVERY trial. EClinicalMedicine. 2023 Dec 6;67:102358. doi: 10.1016/j.eclinm.2023.102358. eCollection 2024 Jan. PMID 38107550
- [Derived] Welzel T, Schobi N, Andre MC, Bailey DGN, Blanchard-Rohner G, Buettcher M, Grazioli S, Koehler H, Perez MH, Truck J, Vanoni F, Zimmermann P, Atkinson A, Sanchez C, Whittaker E, Faust SN, Bielicki JA, Schlapbach LJ; Swissped Recovery Trial. Multicenter Randomized Trial of Methylprednisolone vs. Intravenous Immunoglobulins to Treat the Pediatric Inflammatory Multisystem Syndrome-Temporally Associated With SARS-CoV-2 (PIMS-TS): Protocol of the Swissped RECOVERY Trial. Front Pediatr. 2022 May 20;10:905046. doi: 10.3389/fped.2022.905046. eCollection 2022. PMID 35669398
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT04826588/Prot_SAP_000.pdf